CLINICAL TRIAL: NCT02574364
Title: Abdomen CT and Open Appendicectomy：New Diagnostic and Surgical Procedures
Acronym: ACAOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Municipal No.4 Hospital (Other Government)
Responsible Party: Principal Investigator, weng xinhai, attending physician, Ningbo Municipal No.4 Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: wxinhai
Record Dates: First submitted 2015-09-29; First posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Wound Infection; Complication; Scar
Keywords: abdomen CT; open appendicectomy
MeSH Terms: conditions — Wound Infection; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional incision (Active Comparator): traditional incision : McBurney incision,Rectus incision,Appendix Transverse incision or Tenderness point incision,it was invaginated at the discretion of the surgeon.
  Interventions: Other: traditional incision
- modified incision (Experimental): modified incision :The application of abdomen CT before surgery provides a new approach to the incision and new perception.
  Interventions: Radiation: The application of abdomen CT

INTERVENTIONS:
Radiation: The application of abdomen CT — A modified incision(MI)was designed based on abdomen CT.Using a MI compare traditional incision(TI) to the patient including cut extended, operating time,cut infection, false-positive rate,rehabilitation and return to work.
  Arms: modified incision
Other: traditional incision — McBurney incision,Rectus incision,Appendix Transverse incision or Tenderness point incision,it was invaginated at the discretion of the surgeon.
  Arms: traditional incision

SUMMARY:
The traditional open appendectomy in the clinical effect is not prefect, and for a long time there is no measurable improvement. The application of abdomen CT before surgery provides a new approach to the incision and new perception.

In a randomized controlled trial of modified incision versus traditional incision. Length of hospital day was the primary terminus, while operating time, postoperative complication, scar and time to resume normal activity and work as secondary terminus.

DETAILED DESCRIPTION:
Traditional open appendicectomy have many drawbacks, such as false-positive, cut infection, scar, extended cut, slower rehabilitation and return to work. In the past few years, in order to improve diagnostic accuracy, the abdomen CT is been general applied before appendicectomy, in addition to, a modified incision (MI) was designed based on it. Using a MI compare traditional incision (TI) to the patient including cut extended, operating time, cut infection, false-positive rate, rehabilitation and return to work. It seems that MI would prove superior to TI in terms of hospital day (primary terminus), with operating time, postoperative complication, scar and time to resume normal activity and work as secondary terminus.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical diagnosis of acute appendicitis

Exclusion Criteria:

* children under 14 are not included

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
hospital day | 2 weeks

SECONDARY OUTCOMES:
time to return to normal activity and work in days | up to 4 weeks
operating time in minutes | 180 Minutes
numbers of extended cut, numbers of infection,numbers of intraperitoneal abscess | 1 weeks